CLINICAL TRIAL: NCT03016611
Title: Chewing Ticagrelor Versus Prasugrel in ST-elevation Myocardial Infarction - A Platelet Reactivity Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Elad Asher, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-16-3634
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Acute Coronary Syndrome; STEMI
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing Ticagrelor (Active Comparator)
  Interventions: Drug: Chewing Prasugrel LD
- Chewing Prasugrel (Experimental)
  Interventions: Drug: Chewing Ticagrelor LD

INTERVENTIONS:
Drug: Chewing Ticagrelor LD — 180 mg Chewing Ticagrelor
  Arms: Chewing Prasugrel
Drug: Chewing Prasugrel LD — 60 mg Chewing Prasugrel
  Arms: Chewing Ticagrelor

SUMMARY:
To examine the efficacy of chewing Ticagrelor versus Prasugrel in ST-elevation Myocardial Infarction (STEMI) patients on platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with STEMI
2. Informed, written consent

Exclusion Criteria:

1. Age < 18 years or Age > 75 years
2. Active bleeding; bleeding diathesis; coagulopathy
3. Increased risk of bradycardic events
4. History of gastrointestinal or genitourinary bleeding <2 months
5. Major surgery in the last 6 weeks
6. History of intracranial bleeding or structural abnormalities
7. Suspected aortic dissection
8. Any other condition that may put the patient at risk or influence study results or investigator's opinion (severe hemodynamic instability, unconsciousness, known malignancies or other comorbid conditions with life expectancy <1 year)
9. Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux.
10. Concomitant oral or IV therapy with strong CYP3A inhibitors or strong CYP3A inducers, CYP3A with narrow therapeutic windows
11. Known relevant hematological deviations: Hb <10 g/dl, PLT<100x10^9/l
12. Use of coumadin derivatives within the last 7 days
13. Chronic therapy with ticagrelor, prasugrel, clopidogrel or ticlopidine
14. Known severe liver disease, severe renal failure
15. Known allergy to the study medications
16. Pregnancy
17. Human immunodeficiency virus treatment
18. The use of IIBIIIA receptor antagonists in the 48 hours before enrollment (if abciximab use then in the last 14 days).
19. If the patients cannot sign percutaneous coronary intervention (PCI) informed consent for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Residual platelet reactivity by Platelet Reactivity Units (PRU) VerifyNow 1 hour after Ticagrelor/Prasugrel LD | 1 hour

SECONDARY OUTCOMES:
The percent of patients with a high residual platelet reactivity (PRU > 208) 1 hour, 4-6 hours after Ticagrelor/Prasugrel LD | 4-6 hours
Major, minor, minimal bleeding [ Thrombolysis in Myocardial Infarction (TIMI) criteria] events | 30 days
Occurrence of dyspnea and/or symptomatic bradycardia | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical center, Ramat Gan, Israel